CLINICAL TRIAL: NCT07158944
Title: A Coherent Family Support Model (Co-Fam) for Prevention and Management of Childhood Obesity: Protocol for a Hybrid Type 2 Effectiveness-implementation Trial
Brief Title: Effectiveness of a Family Support Model for Prevention and Management of Overweight and Obesity in Children 6-12 Years
Acronym: Co-Fam
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Liselotte Schäfer Elinder, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01385-01; 2024-02536 (Other Grant/Funding Number: Swedish Research Council); 20230923 (Other Grant/Funding Number: The Swedish Heart Lung Foundation); 20250603 (Other Grant/Funding Number: Stiftelsen Frimurare Barnhuset i Stockholm)
Record Dates: First submitted 2025-08-19; First posted 2025-09-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight
Keywords: Prevention; Obesity treatment; Parental support; Children
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: A hybrid type 2 effectiveness-implementation study will evaluate the effectiveness through a randomized controlled trial with two parallel arms and the implementation through a process evaluation. In addition, a register based control group receiving standard treatment will be collected retrospectively to allow for a national comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives A Healthy School Start and the More and Less program
  Interventions: Behavioral: More and Less
- Control (No Intervention): Receives A Healthy School Start and standard treatment for overweight or obesity

INTERVENTIONS:
Behavioral: More and Less — Dose: 10 group sessions + 6 individual booster sessions Frequency: 10 weekly group sessions (10 weeks) 6 booster sessions every 6th week
  Arms: Intervention

SUMMARY:
The study will evaluate a coherent model of family support including school health care, primary health care and pediatric clinics. The model combines two evidence based programs: the universal "A Healthy School Start" provided to all children and their families during grade 1 and the targeted parental support program "More and Less" provided to parents of children with overweight or obesity.

The hypothesis is that combining the Healthy School Start and More and Less programs in a coherent model will increase the collaboration between regional and municipal stakeholders, ensure early identification of families in need, ultimately improving prevention and treatment of childhood overweight and obesity. The aim of this study is to evaluate the implementation of a coherent model of family support provided through school and primary health care.

DETAILED DESCRIPTION:
In this hybrid type 2 effectiveness-implementation study, a two-armed randomized controlled trial will randomize families to either the intervention arm receiving the More and Less program or the control arm receiving standard care from primary health care or a pediatric clinic. A matched control group will be identified from a national obesity register for supplementary comparison. Eligible participants are families with children aged 6-12 years with overweight or obesity, enrolled in schools implementing the Healthy School Start program. Effectiveness outcomes to evaluate the intervention are BMI z-score, parental feeding practices, diet and physical activity, child eating behaviour and intervention fidelity which will be measured at baseline, three and 12 months. Implementation outcomes will be evaluated in a process evaluation assessing reach, fidelity, acceptability, feasibility and cost, assessed at 12 and 24 months using a mixed methods approach.

ELIGIBILITY:
Inclusion Criteria:

* A parent of a child between 6-12 years of age.
* The child attends a school providing the Healthy School Start program.
* The child has been diagnosed with overweight (age standardized BMI of 25 or above) or obesity (age standardized BMI of 30 or above) by a health care personnel.

Exclusion Criteria:

- If parents are unable to understand and/or communicate in easy Swedish.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
BMI z-score | Measured at baseline, 3 and 12 months.
  The effects on children's BMI z-score (IOTF cut offs) whose parents receive the More and Less program over a 12-month period, compared to children receiving standard treatment

SECONDARY OUTCOMES:
The child's dietary habits | Measured at baseline, 3 and 12 months follow-up
  Assessed using the Eating and Physical Activity Questionnaire (EPAQ).
  Parents are asked to recall the child's intake of unhealthy and healthy foods and unhealthy drinks. Questions are answered as amounts (deciliters, glasses or portions) of 0 to 7 or more. For unhealthy foods - higher numbers are worse, for healthy foods - higher numbers are better.
The child's physical activity level | Measured at baseline, 3 and 12 months
  Assessed through three questions from the Public Health Agency's annual school survey to children, with questions asked to the parents.
  Questions are answered by estimating the number of days a week with physical activity (0-7), number of times a week with exercise (0-7) and time spent sedentary during the week (0-5) - higher numbers are better.
The child's eating behavior | Measured at baseline, 3 and 12 months
  Assessed using the validated Children's Eating Behavior Questionnaire (CEBQ) including 35 questions on eight different scales that help identify behavioral traits that may contribute to obesity or disordered eating and is answered by a parent.
  Answers: Parents rate their child's eating behavior on a five-point Likert scale (never, rarely, sometimes, often, always)
Parental feeding practices | Measured at baseline, 3 and 12 months
  Assessed using the validated Comprehensive Parental Feeding Questionnaire (CPFQ) including five factors: Monitoring of children's food intake, pressure to eat, restriction of food, use of food for emotional regulation, and healthy eating guidance.
  Answers: parents rate their feeding practices on a four-point Likert scale (rarely, sometimes, often, very often) or (disagree, somewhat disagree, somewhat agree, agree).

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte S Elinder, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Primary healthcare, Södertälje, Sweden

IPD SHARING:
Plan to Share IPD: No
The data will not be publicly available due to containing information that could compromise the privacy of the study participants.

REFERENCES:
- See also: Information about the Co-fam study — https://ki.se/en/research/research-areas-centres-and-networks/research-groups/community-nutrition-and-physical-activity-conpa-liselotte-schafer-elinders-research-group/co-fam-co-fam-a-partnership-model-for-health-promotion-and-early-prevention-and-treatment-of-obesity